CLINICAL TRIAL: NCT00575458
Title: Prospective Randomized Comparison of Dynamic Versus Static Splinting After Dupuytren's Contracture Release
Brief Title: Splinting for Dupuytren's Contracture Release
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: David Ring, Massachusetts General Hospital
Other Study IDs: 2005p002466
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Dupuytren's Disease
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Static Splint
- 2: Dynamic Splint

SUMMARY:
This study is comparing two different kinds of splints for patients who have had a surgical contracture release of dupuytren's disease. It compares a static splint and a dynamic splint.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* males and females with Dupuytren's contracture
* patients with contracture of less than 30 degrees of MCP contractions and no contractions of the IP joints

Exclusion Criteria:

* previous surgical treatment for Dupuytren's
* contracture of MCP greater than 30 degrees
* contraindications for dynamic splinting (upper limb amputees, paresis, ect.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orthopaedic Hand Clinic
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2005-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
DASH questionnaire, PCS questionnaire, Wahler Physical Symptom Inventory, CESD questionnaire | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David C. Ring, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States